CLINICAL TRIAL: NCT04244058
Title: Evaluation of Pharmacologically-induced Changes in Excitatory Glutamatergic Neurotransmission of Severe TBI Patients
Brief Title: Changes in Glutamatergic Neurotransmission of Severe TBI Patients
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Given CoVid-19 pandemic we could not recruit subjects/patients for the 1st year. Currently waiting for new sponsor to fulfill the aims.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-09020845
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Disorder of Consciousness; Traumatic Brain Injury
Keywords: Positron emission tomography; 18F-FPEB; NMDA; Dopamine; mGlu5-R; Molecular neuroimaging; Traumatic brain injury; Disorders of consciousness
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries, Traumatic | interventions — Amantadine; Levodopa

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be unaware of the medication used during the pharmacological challenge for the PET approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NMDA blocker (Active Comparator): Comprehensive functional analyses of dynamic [18F]FPEB-PET signal at rest will be carried out in normal volunteers and patients with DOC due to severe brain injury over a 24-month time period. In each study, we will first evaluate mGluR5 occupancy within the frontal cortex, anterior cingulate cortex, insula, striatum and thalamus. Then, a single dose of amantadine (AMT), a compound that blocks NMDA-R and increases glutamate levels at the synaptic cleft, will be given to each subject or patient and at the time corresponding to the peak of the dose, a second [18F]FPEB-PET will be acquired.
  Interventions: Drug: NMDA blocker
- NMDA blocker + L-DOPA (Experimental): All the patients with DOC that participate in ARM 1 will follow the same methodology of ARM 1: measurement of mGluR5 occupancy at rest and following NMDA-R blockade with AMT by means of [18F]FPEB-PET after premedication with L-DOPA introduced 1 hour prior each [18F]FPEB-PET acquisitions.
  Interventions: Drug: Amantadine + L-DOPA

INTERVENTIONS:
Drug: Amantadine + L-DOPA — Amantadine 150 mg L-DOPA 375mg/carbidopa 75mg
  Arms: NMDA blocker + L-DOPA
Drug: NMDA blocker — NMDA blocker
  Arms: NMDA blocker

SUMMARY:
Studies in patients with disorders of consciousness (DOC) after severe brain injury implicate dysfunction of the anterior forebrain mesocircuit dysfunction a key underlying mechanism. The anterior forebrain metabolism in DOC is markedly downregulated across brain regions underpinning highly elaborated cognitive behaviors demonstrating a collapse of the level of synaptic background activity required for consistent goal-directed behavior and arousal regulation. Since dopamine levels are one of the primary controllers of the level of synaptic background activity within these forebrain structures and in regulating excitatory glutamatergic homeostasis, the investigators propose to investigate the specific contribution of presynaptic dopamine function in glutamatergic neurotransmission in posttraumatic DOC. The aim of the present study is to measure metabotropic glutamate receptors 5 occupancy in the main gutamatergic structures of the brain using (3-[18F]fluoro-5-(2-pyridinylethynyl)benzonitrile)-positron emission tomography ( [18F]FPEB-PET) at rest and following a short pharmacological challenge with amantadine, an N-methyl-D-aspartate receptor (NMDA-R) antagonist, following L-DOPA, and amantadine + L-DOPA. Using this novel technique in DOC the investigators will characterize the relevance of a presynaptic deficiency to synthesize and/or release dopamine in the final regulation of excitatory interneurons of the anterior forebrain mesocircuit.

It is unknown whether glutamatergic neurotransmission is affected across the population of subjects with DOC and, if this condition is secondary to a presynaptic dopaminergic failure of the anterior forebrain mesocircuit (i.e., down-regulation). Since the investigators previously identified the existence of a presynaptic dopaminergic deficit in these subjects due to a failure in the biosynthesis of dopamine, the investigators will evaluate if by providing the main biological substrate of the biosynthesis process (i.e., L-DOPA) the glutamatergic system regains homeostasis. The investigators therefore propose to investigate patients with posttraumatic DOC using [18F]FPEB-PET at rest and following short pharmacological challenges aimed at increasing glutamate and dopamine release.

DETAILED DESCRIPTION:
Disorders of consciousness (DOC) produced by severe traumatic brain injuries (TBI) lack systematic evaluation and treatment strategies. Accumulating evidence points to the important and general role of impaired anterior forebrain mesocircuit function following multi-focal brain injuries that produce widespread deafferentation or neuronal cell loss (Schiff, 2010, Fridman et al. 2014). Among important sources of neuromodulation of this mesocircuit, alteration of dopaminergic innervations as a result of impaired biosynthesis of dopamine, neurotransmitter release, or its direct binding to dopamine receptors is implicated as having a critical contribution (Fridman and Schiff, 2014, Giacino et al. 2012). Parallel deficits of long-range excitatory glutamatergic neurotransmission likely play an equally crucial factor in all DOCs (Fridman and Schiff, 2014), as shown in non-human primates where a decrease of cortical glutamate levels occurs following dopamine depletion of substantia nigra (SN), and likely the ventral tegmentum (VT) (Fan et al., 2014). In a Phase 0 clinical trial exploring the pharmacodynamics underlying DOC (NINDS R21-NS093268) the investigators have shown that chronic TBI patients have an underlying presynaptic dopamine deficit in SN and VT that is not reversed by blocking only dopamine reuptake but is reversed by increasing dopamine synthesis using the dopamine precursor L-DOPA (Fridman et al., 2018)*. No prior studies, however, have provided direct measurements of glutamatergic deficits in DOC. Moreover, no systematic evaluation of glutamatergic neurotransmission has been carried in post-TBI DOC patients following dopaminergic modulation. This gap in knowledge is critically important as only one therapeutic intervention has shown modest effectiveness in subacute and chronic stage of TBI (Giacino et al., 2012) targeting glutamatergic neurotransmission without addressing impaired dopaminergic biosynthesis (Fridman et al., 2018)*.

Here the investigators develop a novel and systematic assessment focusing on the role of the integrity of dopaminergic-glutamatergic systems in DOC. The investigators approach allows for evaluation of the integrity of glutamatergic innervations to key neuronal populations within the anterior forebrain mesocircuit. Using a similar approach (i.e., molecular neuroimaging and pharmacological challenges), the investigators have identified that patients with DOC exhibit: 1) a widespread presynaptic deficit affecting the resting dopamine synaptic activity; 2) a widespread presynaptic deficit affecting the induced dopamine release after pharmacological stimulation with amphetamine; and, 3) a partial postsynaptic deficit. The investigators long-term goal is to understand how neuromodulation of the anterior forebrain mesocircuit in DOC can be optimally manipulated for diagnosis and therapy. The investigators working hypothesis is that patients with DOC following TBI have alterations of glutamatergic function that can be partially reversed by dopamine replacement. The rationale that underlies the proposed research is that identification of a glutamatergic down-regulation in DOC as well as identification of the key regulator of this down-regulation (i.e., secondary to a deficit in the synthesis of dopamine) will allow the development of complementary diagnostic methods to predict patients' responses to specific therapies and, further improve the efficacy of neuropharmacological treatments to induce recovery of consciousness following severe TBI by rational polypharmacy. The investigators will develop quantitative measurements to test this hypothesis under the following Specific Aims:

Specific Aim 1a. To identify and characterize impaired glutamatergic neurotransmission deficits in posttraumatic DOC.

The investigators will assess in-vivo the availability of free metabotropic glutamate receptor 5 (mGluR5) at rest in patients with DOC and normal volunteers (NV) following N-methyl-D-aspartate receptor (NMDA-R) blockade with amantadine (AMT) utilizing [18F]FPEB-PET. The investigators working hypothesis is that patients with DOC will demonstrate:

1) a glutamatergic deficit in anterior forebrain mesocircuit that is identified by a lower mGluR5 availability at rest; and 2) a failure to decrease mGluR5 occupancy following stimulation with AMT.

Specific Aim 1b. To determine the reversibility of glutamatergic neurotransmission deficits in response to dopamine replacement in posttraumatic DOC.

In DOC patients with a demonstrated glutamatergic deficit the investigators will assess the availability of free mGluR5 at rest and following NMDA-R blockade with AMT by means of [18F]FPEB-PET after premedication with L-DOPA. The investigators hypothesize that impaired glutamatergic neurotransmission in DOC can be partially restored by providing the dopamine precursor L-DOPA and thus supporting dopamine biosynthesis and subsequent release of a circuit- level inhibition at the level of the thalamus (mesocircuit hypothesis). Impaired biosynthesis is proposed to arise secondary to a posttraumatic enzyme tyrosine hydroxylase deficiency affecting the biosynthesis of dopamine.

The investigators expected outcomes are anticipated to identify biomarkers to better define future therapeutic interventions in TBI patients with DOC. These results are expected to have an important positive impact because the identified biomarkers are highly likely to provide new therapeutic targets to induce recovery and therefore decrease disability and social cost in this large population of severe brain injured patients.

ELIGIBILITY:
Patients Subjects with DOC

Inclusion criteria:

* Age between 18 and 75 years of age, inclusive.
* Patients with disorder of consciousness (vegetative state, minimally conscious state, emerged from minimally conscious state) following severe brain injuries.
* Male or non-pregnant female.
* Medically stable.
* Informed consent from a Legally Authorized Representative.

Exclusion criteria:

* Medical instability.
* Clinical history of moderate to severe hypertension or heart arrhythmia.
* Use of stimulants or dopamine blocker during the 24 hours previous to the study.
* Absence of a legally authorized representative (LAR) to sign the consent form.

Normal Volunteers

Inclusion criteria:

* Age between 18 and 75 years old, inclusive.
* Absence of cardiological, neurological and/or psychiatric diseases.
* Absence of familiar antecedents of sudden death of unknown reason.
* Male or non-pregnant female.
* Informed consent signed.

Exclusion criteria:

- Caffeine or alcohol intake in the last 24 hours previous to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Delta % changes in binding potential nondisplaceable (%ΔBPnd) | Day 1 and Day 2
  BPnd induced by pharmacological challenges using AMT, L-DOPA and, AMT+L-DOPA (%ΔBPnd-AMT, L- DOPA and AMT+L-DOPA, respectively).

SECONDARY OUTCOMES:
Coma Recovery Scale Revised | Day 1 and Day 2
  The Coma Recovery Scale-Revised (CRS-R) is a standardized neurobehavioral assessment measure comprised of six subscales designed to assess arousal level, audition, language comprehension, visuoperceptual, motor function, oromotor capacity, expressive speech, and yes/no communication in patients with disorders of consciousness (DOC).
  The scale comprises 23 items divided into 6 sub-scales. Maximal score is 23 and minimal score is 0, where 0 represents normality and 23 severe coma.

CONTACTS AND LOCATIONS:
Overall Officials: Esteban A Fridman, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will involve a small sample with deficits secondary to traumatic brain injury (i.e., vegetative state and minimally conscious state). These rare disorders are associated with distinguishing features that even with the removal of all identifiers it would be difficult if not impossible to protect the identities of subjects. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
  Data to be share will be 18F-FPEB raw data; CRS-R available data; anatomical data from the MRI.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available from publication date up to 3 years.
Access Criteria: Only under a data-sharing agreement.

REFERENCES:
- [Background] Fridman EA, Osborne JR, Mozley PD, Victor JD, Schiff ND. Presynaptic dopamine deficit in minimally conscious state patients following traumatic brain injury. Brain. 2019 Jul 1;142(7):1887-1893. doi: 10.1093/brain/awz118. PMID 31505542
- [Background] Fridman EA, Schiff ND. Neuromodulation of the conscious state following severe brain injuries. Curr Opin Neurobiol. 2014 Dec;29:172-7. doi: 10.1016/j.conb.2014.09.008. Epub 2014 Oct 3. PMID 25285395
- [Background] Fridman EA, Beattie BJ, Broft A, Laureys S, Schiff ND. Regional cerebral metabolic patterns demonstrate the role of anterior forebrain mesocircuit dysfunction in the severely injured brain. Proc Natl Acad Sci U S A. 2014 Apr 29;111(17):6473-8. doi: 10.1073/pnas.1320969111. Epub 2014 Apr 14. PMID 24733913
- See also: Weill Cornell Medicine Consortium for the Advanced Study of Brain Injury (CASBI) — https://casbi.weill.cornell.edu/